CLINICAL TRIAL: NCT05980923
Title: Thyroid Profiles in Middle Eastern Patients Admitted With Acute Illness: Prevalence, Clinical Features and Impact on Mortality
Brief Title: Thyroid Profiles in Patients With Acute Illness
Status: Withdrawn | Type: Observational
Why Stopped: no funds for TSH testing
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: DCR2023/1.ThyrAcuteIll
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Dysfunction; Acute Illness
Keywords: Thyroid abnormalities; Acute illness; Prognosis; Middle east
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyrotropin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP 1: Acute illness and abnormal thyroid function: Patients admitted to the hospital with acute illness and found to have thyroid function abnormalities.
  Interventions: Other: Performing blood thyroid test (TSH, FT4, FT3)
- GROUP 2: Acute illness and normal thyroid function: Patients admitted to the hospital with acute illness and found to have normal thyroid function.
  Interventions: Other: Performing blood thyroid test (TSH, FT4, FT3)

INTERVENTIONS:
Other: Performing blood thyroid test (TSH, FT4, FT3) — Blood test as above

SUMMARY:
Patients admitted to the hospital with acute illness may have a wide spectrum of thyroid function abnormalities. It is largely unknown whether such aberrations are temporary or persist for a long time, and whether they impact prognosis of such patients.

DETAILED DESCRIPTION:
Recently, there has been a growing body of evidence that subclinical thyroid dysfunction as a contributor to the increase of cardiovascular events. Elevated serum thyroid-stimulating hormone (TSH) levels and normal free thyroxine (FT4) and free triiodothyronine (FT3) levels have been associated with worse heart failure and dyslipidemia. Furthermore, higher risk of atrial fibrillation has been linked tp thyroid abnormalities in these patients.

Patients admitted to the hospital with acute illness may have a wide spectrum of thyroid function abnormalities. It is largely unknown whether such aberrations are temporary or persist for a long time, and whether they impact prognosis of such patients. This study aimed at evaluating the prevalence of thyroid function abnormalities in patients admitted to hospital with acute illness and their temporal changes and impact on mortality during hospitalization and at 1 year. Serum level of thyroid stimulating hormone and free T4 and T3 measured on admission. Clinical and laboratory profiles of patients with abnormal thyroid function (ATF group) will be compared to those with normal thyroid function (NTF group). Short and long term survival of both groups were compares as well.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission
* Adults aged 18 years and above
* Willing to sign an informed consent
* Diagnosis on admission is acute illness that includes: heart failure, acute coronary syndrome, sepsis, acute stroke, hypotension, acute system-organ failure including renal and hepatic failure.

Exclusion Criteria:

* Age less than 18 years.
* Refusal to sign consent.
* Admission for a reason not classified as acute illness.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: nclusion Criteria: All patients admitted to the hospital with acute illness will have their serum level of thyroid stimulating hormone and free T4 and T3 measured on admission. Clinical and laboratory profiles of patients with abnormal thyroid function (Group 1) will be compared to those with normal thyroid function (Group 2). Serum thyroid test will be repeated at 6 months. Short and long term survival of both groups will be compared as well.
  Diagnosis on admission is acute illness includes: heart failure, acute coronary syndrome, sepsis, acute stroke, hypotension, acute system-organ failure including renal and hepatic failure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
In hospital mortality | From time of study entry until the date of death from any cause, assessed up to 2 weeks.
  All-cause death rate in patients with abnormal thyroid function compared with death in those with no abnormal thyroid function during the patients hospital stay..

SECONDARY OUTCOMES:
6-month mortality rate | From date of study entry until the date of death from any cause, assessed up to two weeks.
  All-cause death rate in patients with abnormal thyroid function compared with death in those with no abnormal thyroid function at 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Will contact other ICU physicians in the city of Amman to invite them to participate in the study